CLINICAL TRIAL: NCT03979677
Title: Effects of Lifestyle Modification on Vestibular Migraine
Acronym: LMVM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Richard A. Roberts, Ph.D., Associate Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Vestibular Migraine
Keywords: vestibular migraine, dizziness, vertigo
MeSH Terms: conditions — Dizziness; Vertigo

STUDY DESIGN:
Intervention Model Description: Eligible participants will receive information on food/beverage triggers to avoid, restful sleep tips, simple exercise tips, and eating regularly at the same time. Participants will return after 60 days and both pre- and post-intervention measures will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): All participants will be provided written and verbal instructions regarding the lifestyle modification intervention.
  Interventions: Behavioral: Lifestyle Modifications

INTERVENTIONS:
Behavioral: Lifestyle Modifications — Written suggestions on common migraine triggering food/beverages to avoid, restful sleep tips, exercise suggestions, and eating set mealtimes will be provided as the intervention.

SUMMARY:
Vestibular migraine was recently addressed by the International Headache Society (IHS) as separate from other types of migraine. Vestibular migraine is one of the most common causes of vertigo attacks, affecting 1-5% of people. People with vestibular migraine have lower quality of life compared to others and some are completely debilitated by their symptoms. Symptoms include vertigo, nausea, head motion-induced dizziness, unsteadiness, balance problems, and lightheadedness. Most reports of vestibular migraine management have focused on treatment with medications; however, recommendations also include some form of lifestyle modification. Lifestyle modifications like avoidance of certain foods, improving sleep, exercising, etc. have all been reported to help migraine in general, but there are no reports on the effects of lifestyle modification on vestibular migraine as defined by IHS. It is important to investigate the effects of lifestyle modifications on vestibular migraine because the underlying causes of vestibular migraine are unclear. So, it is also unclear if lifestyle modifications are effective for vestibular migraine. Many investigations of lifestyle modification on migraine include a single modification like diet, weight loss, or sleep. Our modifications include food triggers, restful sleep, exercise, and eating regularity. We hypothesize comprehensive lifestyle modifications will improve symptoms of vestibular migraine. We will measure how people feel dizziness and headache activity is affecting their lives before and after our intervention. This project is important because vestibular migraine is reported to be the one of the most common causes of vertigo and interventions useful for other migraine types may not be effective for vestibular migraine. If we demonstrate improvement with comprehensive lifestyle modifications, we will continue the line of investigation with randomized, controlled studies. This work furthers our goal of helping the many people impacted by vestibular migraine.

DETAILED DESCRIPTION:
Significance Dizziness is a frequently reported symptom encountered by healthcare providers, affecting 20-30% of the general population [9, 10]. Vestibular migraine (VM) is one of the more common causes of dizziness, including rotational vertigo, and is reported to be the diagnosis in 11.4% of patients presenting to specialized dizziness centers [11]. Prevalence ranges between 4.3 - 29.3% depending on diagnostic criteria and population [1]. Clearly, VM affects a large segment of the population presenting with dizziness. It is for this reason that diagnostic criteria for VM were included in the appendix of the beta version of the International Classification of Headache Disorders - 3 (ICHD-3β) [5].

Dizziness Common symptoms with VM include rotary vertigo, positional vertigo, sensitivity to motion, unsteadiness, imbalance, and lightheadedness, among others [1, 2]. These types of symptoms can be debilitating. A recent investigation indicated that nearly 70% of patients with VM rated their symptoms as having a moderate to severe impact on health-related quality of life [3]. The authors used the Dizziness Handicap Inventory (DHI) as a disease-specific subjective measure of health-related quality of life [4].

Headache As one might expect with a form of migraine, headache is common with VM and is included as one of the diagnostic criteria found in ICHD-3β. However, the actual criterion is 50% of episodes associated with at least one of the following: headache, photophobia/phonophobia, or visual aura [5]. This is in keeping with the finding that only about 50% of patients with VM report both headache and dizziness at the same time [12]. It is often the case that the headache is temporally distinct.

Pharmacologic Treatment Treatment of VM has focused primarily on pharmacologic intervention [2, 15]. This is based on the use of this type of intervention for other migraine with and without aura rather than the results of randomized controlled studies in patients with VM [1, 2]. One randomized controlled study found that 38% of patients with VM benefitted from zolmitriptan compared to only 22% benefit in the control group given a placebo [16]. This study only had 8 experimental and 9 control participants. Other investigators have reported 57.6% complete reduction in attack frequency with prophylactic use of various types of medication including propranolol, clonazepam, flunarizine, metoprolol, or amitriptyline [17]. Mikulec et al. found reduction in symptoms for 25% of patients using topiramate and a reduction of symptoms in 46% of patients with nortriptyline [18]. Interestingly, they stated 14% of their patients reported reduced symptoms after eliminating caffeine only from their diets. It is interesting that protocols incorporating some type of lifestyle modification along with pharmacologic intervention seem to report relatively higher overall rates of success, 72% for Reploeg and Goebel [19] and 86-92% for Johnson [20].

Lifestyle Modifications as Treatment We find it noteworthy there was an effect of simple elimination of caffeine reported by Mikulec et al. [18]. As stated above, some investigators included dietary modifications along with pharmacologic intervention. Reploeg and Goebel reported 16% of their patients had complete or well-controlled resolution of their symptoms by dietary modifications alone [19]. They also report the improvement was realized in less than four weeks compared to much longer for patients who went on to need intervention with medication. Although only two investigations specifically reported on dietary triggers alone in VM management, dietary considerations, along with other lifestyle modifications continue to be recommended in published reports of treatment of VM [1, 2]. This is because it is well-known there are various triggers for migraine in general and the assumption is this is also true for VM. Orr [6] provides a thorough review of the effects of diet interventions on migraine in general. For diets attempting to eliminate triggering food/drink, the results suggest significant reduction of migraine symptoms in a range of 63-93% of participants. The results of diet modification alone are at least as compelling compared to the results reported for many types of medication. Restful sleep is another factor that seems to improve symptoms of migraine. Smitherman et al. [8] used cognitive behavioral therapy to treat insomnia, a common comorbid symptom reported in migraineurs. They found a 48.9% reduction of headache frequency for the experimental group compared to the control group (25%) at six weeks follow-up. These authors point out another interesting influence on migraine. Their control group actually did experience reduction in headache frequency even without intervention for insomnia. Smitherman et al. related this to their "sham" control that actually may have helped regulate eating times for these participants. Missing meals or fasting is a trigger in as many as 57% of migraineurs [21]. Dieterich et al., in their review of VM treatment, mention the positive effects of vestibular rehabilitation therapy on reduction of migraine [2]. They point out that physical activity, in general, has some benefit on migraine. So, the assumption is that it is the associated adaptation and substitution that is helpful with VRT. In fact, it could just be increased activity. Varkey et al. [22] note a linear relationship between low physical activity and frequency of migraine in general. By increasing physical activity through exercise, it has been suggested that a 40% reduction in migraine headache frequency can be realized [7]. This has not been studied in VM. In fact, there are no specific investigations on the effects of individual lifestyle modifications, much less comprehensive lifestyle modifications, on VM. Two investigations have some data showing modest improvement with slight modification, not comprehensive lifestyle modifications [18, 19].

In the current project we hypothesize that comprehensive lifestyle modifications chosen to decrease migraine activity will be effective at reducing symptoms of vestibular migraine.

Innovation Previous studies have shown that pharmacologic intervention can be effective for management of VM, but participant groups were not homogeneous and results are variable. Studies incorporating pharmacologic intervention plus diet restrictions also seem effective but with variable results. Studies of patients with VM that have used isolated dietary restrictions with no pharmacologic intervention indicate modest improvement. The current project is innovative in at least two ways. First, we will use a comprehensive lifestyle modification approach with control of dietary triggers, improvement in restful sleep, increased physical activity, and eating on a regular daily schedule. All of these management approaches have shown promise in improving symptoms in patients with migraine in general but have not been combined into a single intervention in patients with vestibular migraine. Second, we will have a more homogeneous participant group by using the ICDH3β criteria to diagnose vestibular migraine. This is a likely source of variability in the other published work on treatment of vestibular migraine. There was not consensus on these criteria until more recently. The proposed investigation has the potential to improve the way patients with VM are managed. It is also possible that our results will help other researchers in their efforts to determine the cause of VM.

Research Plan We propose to test the hypothesis that comprehensive lifestyle modifications will improve symptoms of vestibular migraine. Previous investigations using pharmacologic intervention are variable in terms of results and range from 25-100% control of VM symptoms. Some of these reports were retrospective and many had a small sample size. Interestingly, the reports that included both some form of lifestyle modification along with pharmacologic intervention had less variable results (72-92%). This is interesting because the effects of lifestyle modification without pharmacologic intervention on migraine, in general, seem promising (63-93% control with diet; 48.9% control with improved sleep; 40% control with exercise; and even 25% control with regular eating times). This compares well to the results with either pharmacologic intervention alone or pharmacologic plus dietary intervention. This evidence forms the basis for our hypothesis.

Specific Aim. Determine the effects of comprehensive lifestyle modifications on subjective measures of the impact of vestibular migraine on health-related quality of life.

Hypothesis. Comprehensive lifestyle modifications will improve self-perceived impact of the symptoms of dizziness and headache in individuals with vestibular migraine.

Rationale There is ample evidence in the literature on treatment of migraine, in general, that lifestyle modifications can improve patient status. This is true for elimination of food/drink triggers, improved sleep, improved exercise habits, and consistency with eating times. Even though lifestyle modifications are sometimes included in guidelines on treatment of VM, there is only little evidence in the literature and this relates to elimination of caffeine only or triggering food/drink. Those studies showed modest effects even though the effects of lifestyle modification on migraine in general are much greater and approach 93% control of symptoms. We hypothesize that by using a comprehensive lifestyle modification regimen, there will be a greater improvement in patient outcome than what has been reported for vestibular migraine with caffeine only or food/drink trigger elimination only which improved 14-16% of their participants. This hypothesis will be tested by obtaining pre-treatment and post-treatment measures.

Experimental Approach All patients presenting for evaluation of dizziness and imbalance at our facility who meet the criteria for vestibular migraine as defined by ICHD-3β will be offered the opportunity to participate in this investigation. Regarding sample size, this is a preliminary study. Other investigations of VM intervention have used sample sizes ranging from 5 participants to 111 participants. We have chosen a sample size of 40 for this preliminary investigation.

1. Properly consented participants will complete the DHI and the HDI. These pre-treatment scores will be used as a measure of the effects of vestibular migraine on dizziness and headache impact on health-related quality of life. Participants will also use a 5-point Likert scale to rate their agreement with statements about current ingestion of common migraine triggers, restful sleep, exercise, and regularity of eating schedule.
2. Participants will be instructed in our comprehensive lifestyle modification program. Information will be presented verbally and in written format for later participant reference. Participants will be instructed to refrain from all common food/drink triggers for migraine. Participants will receive information on improving sleep hygiene to enhance restful sleep. Participants will be encouraged to exercise at the same time daily. Participants will be counseled to eat at the same times during the day.
3. Participants will be compensated with a $25 gift card at this point in the investigation (Pending VICTR funding).
4. Participants will commit to the comprehensive lifestyle modification plan for 60-days. It has been reported that when lifestyle modifications were effective in VM, the response took less than four weeks. 60-days encompasses that duration but also may allow for future comparison with pharmacologic studies which need a longer time for an effect.
5. The study endpoint for each participant will be after 60-days on the comprehensive lifestyle modification plan. At that time, participants will return to the Balance Disorders Laboratory and complete post-treatment DHI and HDI, as well as their agreement with the Likert scale statements. Finally, participants will be asked to rate their perceived compliance with each parameter of the comprehensive lifestyle modification plan.

7. Participants completing the post-treatment measures will receive another $25 gift card in compensation (Pending VICTR funding).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older)
* Must meet International Classification of Headache Disorders criteria for vestibular migraine
* Must be able to read and comprehend the English language as instructions are only provided in that language

Exclusion Criteria:

* Younger than 18 years
* Do not meet IHCD criteria for vestibular migraine
* Unable to understand English language instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts RA, Watford KE, Picou EM, Hatton K, Trone TH, Brignola EY. Effects of Lifestyle Modification on Vestibular Migraine. Otol Neurotol. 2021 Dec 1;42(10):e1537-e1543. doi: 10.1097/MAO.0000000000003297. PMID 34325453

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Lifestyle Modification Intervention Group: Participants were recruited from patients seen for consultation for dizziness and/or imbalance in the John S. Odess Otolaryngology and Head and Neck Surgery Clinic. Consultations were provided by two nurse practitioners and one otolaryngologist. All clinicians were experienced in diagnosis and management of dizziness and imbalance including VM. All adult patients diagnosed with definite VM using the consensus criteria4 were eligible for inclusion. Patients who were determined to need pharmacological management at initial consultation were excluded.
Period: Overall Study
Arm/Group | Single Lifestyle Modification Intervention Group
Started | 41 (Participants enrolled)
Completed | 28 (participants completed)
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Single Lifestyle Modification Intervention Group
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Headache Disability Inventory (HDI)
Description: This measure assesses disease-specific (headache) health-related quality of life using a 0 - 100 scale with 0 indicative of no impact and 100 indicative of severe maximum impact. We will assess change in HDI score by comparing baseline performance to performance 60-days after intervention.
Time Frame: Change in HDI total score will be determined 60-days post intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 28
score on a scale | 14.3 [8.94 to 19.67]
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other — HDI and DHI analyzed using linear mixed-effects models with two within-participant factors, Intervention (pre-intervention, post-intervention) and Inventory (DHI, HDI). All models included participant as a random factor. Models constructed using lmer function of the lme package in R and analyzed using anova function in base R. Significant main effects and interactions were evaluated using emmeans . Pairwise comparisons were adjusted to account for false-discovery rates; p < .0001, linear mixed-effects models — Multiple comparisons were adjusted

2. Primary Outcome: Dizziness Handicap Inventory (DHI)
Description: This measure assesses disease-specific (dizziness) health-related quality of life using a 0 - 100 scale with 0 indicative of no impact and 100 indicative of severe maximum impact.We will assess change in DHI score by comparing baseline performance to performance 60-days post-intervention.
Time Frame: Change in DHI total score will be determined 60-days post intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 28
score on a scale | 14.3 [8.94 to 19.67]
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p < .0001, linear mixed-effects models — Point change in DHI was tests

ADVERSE EVENTS:
Time Frame: 105 days, SD = 78 days
Arm/Group | Single Lifestyle Modification Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
The current study is limited by lack of a control group. Future investigations could incorporate crossover interventions to compare effects of no intervention to lifestyle modification, pharmacological intervention, and combinations. Another limitation is that we relied solely on patient report to determine intervention compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT03979677/Prot_SAP_ICF_000.pdf